CLINICAL TRIAL: NCT02422212
Title: Diet-induced Thermogenesis in Patients With Postoperative RYGBP Weight Regain
Brief Title: Diet-induced Thermogenesis in Patients With Postoperative Roux-in-Y Gastric Bypass (RYGBP) Weight Regain
Acronym: RYGBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Silvia Leite Faria (Other)
Collaborators: University of Brasilia (Other)
Responsible Party: Sponsor-Investigator, Silvia Leite Faria, Ph D, Gastrocirurgia, Brazil
Organization: Gastrocirurgia, Brazil (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 05
Record Dates: First submitted 2015-04-09; First posted 2015-04-21 (Estimated); Last update posted 2015-04-23 (Estimated); Status verified 2015-04

CONDITIONS: Obesity; Bariatric Surgery Candidate; Protein-energy; Imbalance
Keywords: metabolism; Diet Induced Thermogenesis; weight regain; energy expenditure; bariatric
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- healthy weight group (Active Comparator): Postop RYGBP patients who underwent surgery at least 2 years previously and have healthy weight (at least 50% loss of excess weight) (HW group) Intervention: Immediately after RMR measurement, a solid mixed meal was served (270 kcal: 62% carbohydrate, 12% protein and 26% lipid)
  Interventions: Other: patients eat a mixed solid meal
- Obese group (Other): Clinically severe obese patients (Body Mass Index greater than 40 kg/m2, without co-morbidities and greater than 35 kg/m2 with co-morbidities) (OB group) Intervention: Immediately after RMR measurement, a solid mixed meal was served (270 kcal: 62% carbohydrate, 12% protein and 26% lipid)
  Interventions: Other: patients eat a mixed solid meal
- weight regain group (Active Comparator): Patients who suffered weight regain after RYGBP (at least 10% above the minimum weight after surgery and less than 50% loss of preop excess weight) (WR group) Intervention: Immediately after RMR measurement, a solid mixed meal was served (270 kcal: 62% carbohydrate, 12% protein and 26% lipid)
  Interventions: Other: patients eat a mixed solid meal

INTERVENTIONS:
Other: patients eat a mixed solid meal — The three groups were given an indirect calorimetry examination to measure their resting metabolic rate (RMR), respiratory exchange rate (RER) and DIT. The patients collected urine during 24 hours for urinary nitrogen analysis. Immediately after the RMR measurement, patients received a solid mixed meal (270 kcal, with 62% carbohydrate, 12% protein and 26% lipid). Ten minutes after beginning this food intake, postprandial (PP) energy expenditure measurements were taken in the following sequences (in minutes): 10-20, 20-30, 30-40, 60-70, 70-80, 80-90, 110-120, 120- 130, 130-140, 160-170 and 170-180.The DIT was calculated for each time interval.

SUMMARY:
Introduction: According to the National Health and Nutrition Examination Survey 2009-2010, 78 million American adults are obese. Bariatric surgery can provide for a sustained long-term weight loss and the metabolic change caused by the surgery seems to be the main cause of this loss. Cross-sectional, prospective and experimental studies, carried out during the post-operative period of Roux-en-Y Gastric Bypass surgery (RYGBP) have shown an increase of over 200% in energy expenditure after meals Diet-induced Thermogenesis (DIT), a specific component of energy expenditure) when compared with obese patients. However, despite this metabolic improvement, 20-50% of the patients can suffer weight regain about 2 years after surgery. So one question whether such metabolic benefits remain active following post-operative weight regain, or if the disappearance or decrease of these metabolic benefits may be seen as causes of this weight regain.

Objective:To evaluate whether there are DIT differences between patients who maintained weight loss and those who regained weight in the late postoperative (postop) period of RYGBP and those who continue with preoperative (preop) obesity.

DETAILED DESCRIPTION:
Methods: This cross-sectional study evaluated three female groups: 1) Postop RYGBP patients operated at least 2 years previously, with healthy weight (at least 50% loss of excess weight) - HW group ; 2) Clinically severe obese patients (BMI > 40 kg/m2, without co-morbidities or > 35 kg/m2 with co-morbidities) - OB group; 3) Post-op RYGBP WR patients (at least 10% above post-op minimum weight and less than 50% loss of preop excess weight) - WR group. All patients, from a private practice in Brasilia, were given indirect calorimetry examinations (GERATHERM RESPIRATORY®) measuring resting metabolic rate (RMR), respiratory exchange rate (RER) and DIT and collected urine during 24 hours for analysis. Immediately after RMR measurement, a solid mixed meal was served (270 kcal: 62% carbohydrate, 12% protein and 26% lipid). Remove? After ten minutes, successive PP energy expenditure measurements were taken (after some minutes, viz): 10-20, 20-30, 30-40, 60-70, 70-80, 80-90, 110-120, 120- 130, 130-140, 160-170 and 170-180, accompanying a 3-hour measurement period. DIT, calculated for each interval, followed this equation: DIT = PP Metabolic rate (MR) time interval - RMR. Correct? Mean areas under the curve (AUC) of all groups and baseline time measurements were compared using the analysis of variance test (ANOVA). Between-group longitudinal changes were tested using a mixed-effects model analysis of variance for repeated measures. Showing a p-value < 0.05, a Bonferroni correction was used. AUC was calculated by trapezoidal rule, considering significant a value of p <0.05.

Results: 45 patients participated (HW 21, OB 13, WR 11). Mean group age was 37.00 ± 6.98 years , 38.72 ± 7.01 years, and 37.88 ± 6.39 years, respectively. I changed the sequence to match the original. RER values increased significantly in all groups from baseline until final measurements. Metabolic rate (MR) adjusted for body weight (BW-adjusted MR (MR/kg)?) was not significant in the OB group at any PP moment compared to baseline. The HW and WR groups showed significant increase until final measurements. Mean AUC values for RER and RMR in absolute terms did not differ between groups (p = 0.3111 and p = 0.1131, respectively). (Two p values for how many groups ? 2 or 3?) Mean AUC values for BW-adjusted MR (kcal/kg)? differed between groups, where the average AUC value was significantly greater in the HW group than in the WR and the OB groups (p <0.0001 for both). Mean AUC value for BW-adjusted MR in the WR group was not significantly different from the OB group (p = 0.6369).

ELIGIBILITY:
Inclusion Criteria:

* Bariatric patients (those who had done Roux-en-Y Gastric Bypass) who have more than 2 years of surgery with healthy weight and also those with weight regain
* Obese population in pre operative phase of bariatric surgery

Exclusion Criteria:

* Patients if male sex,
* pregnant or breastfeeding patients,
* patients with more than 5 years of surgery

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-01; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Measurement of Diet Induced thermogenesis | 180 minuts
  The three groups were given an indirect calorimetry examination (GERATHERM RESPIRATORY®) to measure their resting metabolic rate (RMR), respiratory exchange rate (RER) and DIT. To assure proper measurement of RER, the patients collected urine during 24 hours for urinary nitrogen analysis. Immediately after the RMR measurement, patients received a solid mixed meal of 270 kcal, which was 62% carbohydrate, 12% protein and 26% lipid. Ten minutes after beginning this food intake, postprandial (PP) energy expenditure measurements were taken in the following sequences (in minutes): 10-20, 20-30, 30-40, 60-70, 70-80, 80-90, 110-120, 120- 130, 130-140, 160-170 and 170-180. In this way, a PP-time period of 3 hours was accompanied. The DIT was calculated for each time interval, based on the following equation: DIT = Metabolic rate (MR) PP time interval as X - RMR.

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Gastrocirurgia de Brasilia, Brasília, Federal District
  - Gastrocirurgia, Brasília, Federal District

REFERENCES:
- [Background] Faria SL, Faria OP, Cardeal Mde A, Ito MK, Buffington C. Diet-induced thermogenesis and respiratory quotient after Roux-en-Y gastric bypass surgery: a prospective study. Surg Obes Relat Dis. 2014 Jan-Feb;10(1):138-43. doi: 10.1016/j.soard.2013.09.020. Epub 2013 Oct 10. PMID 24507080
- [Background] Faria SL, Faria OP, Cardeal Mde A, de Gouvea HR, Buffington C. Diet-induced thermogenesis and respiratory quotient after Roux-en-Y gastric bypass. Surg Obes Relat Dis. 2012 Nov-Dec;8(6):797-802. doi: 10.1016/j.soard.2012.06.008. Epub 2012 Jul 23. PMID 22884301
- [Background] Stylopoulos N, Hoppin AG, Kaplan LM. Roux-en-Y gastric bypass enhances energy expenditure and extends lifespan in diet-induced obese rats. Obesity (Silver Spring). 2009 Oct;17(10):1839-47. doi: 10.1038/oby.2009.207. Epub 2009 Jun 25. PMID 19556976